CLINICAL TRIAL: NCT05855694
Title: Pilot Study of Photobiomodulation for Cancer-Related Cognitive Impairment
Brief Title: Photobiomodulation for Cancer-Related Cognitive Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arash Asher, MD (Other)
Collaborators: Thor (Unknown)
Responsible Party: Sponsor-Investigator, Arash Asher, MD, Director, Cancer Survivorship and Rehabilitation, Patient and Family Support Program, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IIT2022-14-ASHER-HELMET
Record Dates: First submitted 2023-05-04; First posted 2023-05-11 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cancer-related Cognitive Impairment
Keywords: Cancer Survivor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention Arm - Therapeutic Setting (Experimental): Photobiomodulation Helmet, Therapeutic setting, 35mW/cm2 = 42J/cm2, 3 x Sessions per week for 6 weeks
  Interventions: Device: THOR LED Photobiomodulation Helmet - Therapeutic
- Control Arm - Non-Therapeutic Setting (Sham Comparator): Photobiomodulation Helmet, Non-Therapeutic setting, 0mW/cm cm2 = 0J/cm2, 3 x Sessions per week for 6 weeks
  Interventions: Device: THOR LED Photobiomodulation Helmet - Control

INTERVENTIONS:
Device: THOR LED Photobiomodulation Helmet - Therapeutic — Photobiomodulation (PBM) is a non-invasive treatment option that uses nonionizing light sources such as laser diodes and light-emitting diodes in the visible and near-infrared spectrum.
  Each participant will be required to sit with the helmet device over their head for the length of their study session. Participants and study staff will wear protective goggles throughout each session. These goggles help to block out any red LED light emitted from the helmet device. Participants may experience a pleasant warmth upon their head during both the therapeutic and control settings.
  Helmet will be in 'therapeutic setting' of 35mW/cm2 = 42J/cm2
  Arms: Intervention Arm - Therapeutic Setting
Device: THOR LED Photobiomodulation Helmet - Control — Each participant will be required to sit with the helmet device over their head for the length of their study session. Participants and study staff will wear protective goggles throughout each session. These goggles help to block out any red LED light emitted from the helmet device. Participants may experience a pleasant warmth upon their head during both the therapeutic and control settings.
  Helmet will be in 'non-therapeutic setting' of 0mW/cm2 = 0J/cm2
  Arms: Control Arm - Non-Therapeutic Setting

SUMMARY:
This is a single site, pilot randomized, double blinded control trial designed to assess changes in cognitive symptoms in cancer survivors with cancer-related cognitive impairment. Patients will be randomized into one of two Arms: Intervention or Control.

* Arm A: Intervention Group: Use of the THOR LED Photobiomodulation helmet 3x per week for 6 weeks. Helmet will be in 'therapeutic setting', 35mW/cm2 = 42J/cm2
* Arm B: Control Group: Use of the THOR LED Photobiomodulation helmet 3x per week for 6 weeks. Helmet will be in 'placebo setting', 0mW/cm2 = 0J/cm2

This study has been designed to assess the hypothesis that Photobiomodulation can have a positive impact on cognitive symptoms in cancer survivors with cancer-related cognitive impairment.

30 participants will be recruited for this study, 15 per group. Self-report questionnaires assessing cognitive concerns, cognitive abilities, quality of life, depression, and anxiety will be administered at three timepoints through the study Baseline, End of Study Visit and 1 Month Follow Up

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* Previous diagnosis of stage I-III non-central nervous system solid tumor malignancy, Hodgkin, or Non-Hodgkin lymphoma
* Completed cancer treatment (chemotherapy and/or radiation) more than 6 months ago but less than 5 years ago (Current concurrent endocrine therapy, anti-HER-2 therapy allowed, or other stable maintenance therapies (such as rituximab) will be allowed.
* Self-reported cognitive complaints (score ≤ 54 on the Functional Assessment of Cancer Therapy-Cognition, Version 3, Perceived Cognitive Impairment subscale)
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Ability to read, write and understand either English OR Spanish.

Exclusion Criteria:

* Current pregnancy or nursing status
* Current use of Photobiomodulation (PBM) (for any reason)
* A lifetime history of any brain tumor or central nervous system metastasis
* Previous use of intrathecal chemotherapy, chimeric antigen receptor treatment (CAR-T), or stem cell/marrow transplant
* Known history of other neurological conditions involving impaired cognitive function (such as Alzheimer's Disease and related dementias, Parkinson's Disease, or Multiple Sclerosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Cognitive Symptoms | 1-Month Follow Up
  Cognitive symptoms will be measured by changes in scores on the PROMIS Cognitive Function-Short-Form 8a. Scores can range from 8-40. with higher score representing better outcomes.

SECONDARY OUTCOMES:
Cognitive Abilities | 1-Month Follow Up
  Cognitive Abilities will be measured by changes in scores in the PROMIS Cognitive Function Abilities - Short Form 8a. Scores can range from 8-40. with higher score representing better outcomes.
Quality of Life | 1-Month Follow Up
  Quality of Life will be measured by changes in scores the PROMIS-29. Scores can range from 30-140, with higher score representing better outcomes.
Depression | 1-Month Follow Up
  Depression will be measured by changes in scores the PROMIS-29. Scores can range from 4-20, with higher score representing better outcomes.
Anxiety | 1-Month Follow Up
  Depression will be measured by changes in scores the PROMIS-29. Scores can range from 4-20. with higher score representing better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Arash Asher, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Clinical Trial Recruitment Navigator, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No